CLINICAL TRIAL: NCT06767358
Title: Ketamine Sedation in the Intensive Care Unit: a Pilot Randomized Controlled Trial
Brief Title: Ketamine Sedation in the ICU (KANINE) RCT
Acronym: KANINE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 202405KTMN
Record Dates: First submitted 2024-12-11; First posted 2025-01-09 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Mechanical Ventilation; Critically Ill Intensive Care Unit Patients
Keywords: sedation; mechanical ventilation; intensive care unit; critically ill
MeSH Terms: conditions — Critical Illness | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: This RCT plans to study the use of an adjunctive ketamine infusion versus placebo in critically ill mechanically ventilated patients.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine (Experimental): Continuous ketamine infusion (0.50 mg/kg/hour)
  Interventions: Drug: ketamine hydrochloride
- Placebo (Placebo Comparator): Normal Saline Placebo
  Interventions: Other: Normal saline placebo

INTERVENTIONS:
Drug: ketamine hydrochloride — Continuous adjunctive ketamine infusion at a fixed dose of 0.50mg/kg/hour
  Arms: Ketamine
Other: Normal saline placebo — Normal saline placebo infusion
  Arms: Placebo

SUMMARY:
Sedation is given to intensive care unit (ICU) patients to treat discomfort, anxiety, agitation, and to help facilitate care, particularly when they require a breathing tube. Sedation is very commonly used in the ICU with North American data showing almost 40% of ICU patients get sedation to help when they are requiring a breathing machine. Various medications can be given intravenously to provide sedation in the ICU but there are side-effects associated with each such as decreasing a patient's own drive to breathe, and delirium or acute confusion, both of which are associated with worse outcomes. Also, most drugs used for sedation don't treat pain. As a result, many ICU patients are also given narcotics for pain control which can result in tolerance, dependence, and withdrawal. Ketamine is a sedating medication that also treats pain and is often used in the Emergency Department and in the Operating Room but for whatever reason is not commonly used in the ICU.

The investigators are proposing a study to examine the usefulness and safety of adding an intravenous infusion of ketamine to usual care in adult patients that are on a breathing machine in the ICU.

Study Methods The KANINE study is being done at hospitals across Ontario, Canada. It is a randomized controlled trial which means patients will be randomized (akin to a coin flip) to receive ketamine or usual care without ketamine. The study will be blinded which means that neither patients or the doctors will know if the patient is getting ketamine or not, those that get randomized to usual care without ketamine will get an intravenous solution that looks the same as the ketamine infusion. This is important to make sure the results aren't biased in any way. The investigators will include adult ICU patients on a breathing machine who are early in their ICU admission. As most patients will be unconscious, the investigators will ask substitute decision makers (families or caregivers) of patients for informed consent prior to the study commencing. Regardless of whether patients get randomized to ketamine or not, the investigators will make sure that all patients will be adequately sedated and have their pain managed as per usual care.

Setting This study will be performed in adult ICUs across Canada.

Population The investigators will include adults admitted to the ICU on a breathing machine and expected to remain mechanically ventilated beyond the calendar day after randomization. The investigators will exclude patients if: (i) they were admitted with a brain bleed, traumatic brain injury, or stroke; (ii) Admitted with uncontrolled high blood pressure; (iii) admitted with status asthmaticus; (iv); admitted to the ICU with partial thickness burns greater than 10% total body surface area or any full thickness burns; (v) if they have a history of schizophrenia; (vi) if they have very bad liver failure; (vii) if they are palliative or only for comfort care; (viii) if they are requiring very high doses of blood pressure support medication to increase their blood pressure; (ix) if they are receiving a medication that causes paralysis, sometimes used in patients with very bad lung disease; (x) if they have a tracheostomy which means a whole in their neck that they breathe through; (xi) if they are allergic to ketamine; (xii) if they've had a liver transplant in the last month; (xiii) if they are pregnant or breast-feeding.

Outcomes The investigators will follow all the study patients to see if their outcomes are different depending on whether they get randomized to ketamine or not. The investigators will capture how much time they are on the breathing machine, whether they survive or die, how long they stay in the ICU and whether they require a tracheostomy which is a procedure often done on patients who require the breathing machine over a prolonged period of time.

The investigators will also capture how often they get delirious and for those that get delirious how long it lasts for. The investigators will capture how much of other sedating medications study patients use such as antipsychotics and benzodiazepines. The investigators will capture outcomes such as how often study patients get post-traumatic stress disorder after leaving the ICU and how well their pain relief is addressed during their ICU stay. Finally, the investigators will capture side effects related to ketamine or other sedating drug use.

DETAILED DESCRIPTION:
Research question for the KANINE Pilot RCT Is it feasible to perform a larger RCT in mechanically ventilated adult critically ill patients requiring sedation to investigate whether an adjunctive ketamine infusion versus placebo improves patient important outcomes?

Pilot Study Design & Study Centers This is a multi-centre, stratified, allocation-concealed, blinded parallel-group pilot RCT. The primary outcome for this pilot trial will be feasibility as assessed by three outcomes of consent rate, recruitment rate, and protocol adherence. The investigators plan to enroll patients at 4 study centers which are all academic teaching hospitals in Ontario (St Joseph's Hospital, Mount Sinai Hospital, Juravinski Hospital, and the Hamilton General Hospital).

Informed Consent When an eligible patient is identified, research coordinators will approach the patient's SDM a priori to explain the objectives of the trial along with its potential risks and benefits. The informed consent will also include the study protocol description, potential benefits, expected length of the study, and the option to withdraw from the study at any time. The investigators have submitted our REB application to Clinical Trials Ontario and are the final stages of ethics approval.

Allocation & Randomization Once the research coordinators have identified a potentially eligible patient, they will log into our centralized data center. Once connected, computerized prompts will be given for preliminary identifying data. If eligibility criteria are met, a priori consent will be obtained and the patient will be randomly allocated in a 1:1 ratio to either adjunctive ketamine or placebo. Randomization will be stratified by site.

Experimental & Control Interventions All eligible patients assigned to the treatment group will receive an adjunctive ketamine infusion at a fixed dose of 0.50 mg/kg/hour. This will be added to the existing sedative and/or analgesic regime that was selected by the bedside clinician (e.g., propofol and/or midazolam and/or dexmedetomidine and/or fentanyl). The dosing of the first-line sedative and/or analgesic infusion will be titrated to achieve the desired Richmond Agitation Sedation Scale (RASS) at the discretion of the healthcare team rather than titrating the fixed dose ketamine.

If the patient's RASS is lower than the goal, the first-line sedative drug will be titrated down. If the goal RASS has still not been achieved after the first-line sedative agent has been titrated all the way down and stopped, it is suggested that any other additional sedative infusion also be titrated down and stopped. If the goal RASS has still not been achieved, the study drug may be discontinued or held at the discretion of the healthcare team. If the RASS remains lower than the goal, the healthcare team will re-assess the patient to rule out other causes for their decreased level of consciousness. The healthcare team can subsequently resume the study drug infusion if they wish to keep the patient sedated. If the patient's RASS is higher than the goal, the first-line sedative drug will be titrated up as needed at the direction of the healthcare team. If the goal RASS has still not been achieved after the first-line sedative agent has been optimized (based on the discretion of the healthcare team), the study drug dose will not be adjusted and instead, the healthcare team may consider boluses of the primary sedative agent or a third non-ketamine sedative or analgesic infusion.

Unless meeting pre-specified stopping criteria, the study drug will continue for a maximum of 14 days or until the patient is extubated, has undergone a tracheostomy, or has died, whichever occurs first. If patients are re-intubated during the same ICU admission, they will resume the trial and study drug. The maximum duration of the study drug of 14 days will begin on the first day of enrolment (i.e. if a study drug is held for 2 days, the total duration of the patient being exposed to the study drug will still be 14 days from the initiation of the study drug meaning that the patient will not receive the study drug for an additional 2 days to account for the days they were not exposed to it). Conversely, if patients are or re-admitted to the ICU, they will not be eligible to resume the trial nor study drug. However, if a patient remains intubated after their first-line sedation and the study drug have been weaned off, and they need to resume sedatives, the study drug can be restarted. Study drug will continue for 14 days maximum as most intubated patients at that point in time have either been extubated or transitioned to a tracheostomy. If a patient undergoes a tracheostomy during their index ICU stay, the study drug will stop. Furthermore, all enrolled patients will have their liver enzymes tested weekly, or more frequently at the clinician's discretion.

Open-label continuous infusion ketamine will be disallowed while the patient is receiving the study drug. If open-label continuous infusion ketamine is used in this circumstance, it will be considered and recorded as a protocol violation. Open-label bolus ketamine will be allowed in the study.

Control Interventions Patients randomized to placebo will receive normal saline in a 150 mL bag that will look identical to the ketamine infusion. Healthcare providers will follow the same sedation titration chart outlined in Figure 3 and in the Experimental Interventions section. The investigators will disallow open-label continuous infusion ketamine use in both treatment groups.

If the healthcare team chooses to use an open-label continuous ketamine infusion as part of their treatment plan, the study drug would be held in that circumstance until the open-label continuous ketamine had been stopped. If the healthcare team chooses to use open-label bolus dosing of ketamine, the study drug would continue.

Blinding Patient allocation will be blinded to treating physicians, nurses, patients, the biostatisticians associated with the study, site investigators, and the research coordinators collecting the data.

Outcomes

Pilot Study Primary Feasibility Outcomes The primary outcome for the KANINE Pilot Trial is feasibility, which will be judged by 3 outcomes of recruitment rate, consent rate, and protocol adherence.

Recruitment rate:

The investigators define a successful recruitment rate of 0.5 patients per centre per month over the duration of the trial (or 2 patients per month overall across the 4 centres).

Consent rate:

The investigators will define >75% consent rate as successful.

Protocol adherence:

The investigators will define ≥75% protocol adherence as successful

Pilot Study Secondary Clinical Outcomes Ventilator-free days at 28 days, 28-day mortality, ICU mortality, ICU length of stay, tracheostomy, hospital mortality, hospital length of stay, delirium (using the validated Confusion Assessment Method for the ICU (CAM-ICU) score or Intensive Care Delirium Screening Checklist), delirium-free/coma-free days at 14 days, use of antipsychotics (total dosage), use of benzodiazepines (total dosage), post-traumatic stress disorder symptoms at 3 months post-ICU discharge using the validated Impact of Event Scale-Revised, continuous sedative and analgesic requirements over ICU stay, adverse events (arrhythmias, vomiting).

Pilot Study Data Collection Trained research coordinators at each site will screen and log patients admitted to the ICU daily. They will record the following on pre-established data abstraction forms that will be transcribed into a web-based case report form on REDCap Coud that will be encrypted and password protected. The online database the investigators plan to use fully complies with FDA and Health Canada rules for electronic data management.

Statistical Analysis

Sample Size The sample size for the pilot was calculated using a 95% confidence interval approach for protocol adherence. Protocol adherence is defined as: (i) not receiving open-label ketamine for patients in the control arm; and (ii) receiving ketamine for patients in the intervention arm. The lower bound for the confidence interval was set at the threshold for feasibility (75%) and an expected adherence rate (90%) was selected based on a previously published RCT24. Using a power of 80%, the require sample size is at least 48 patients. To be conservative, the investgiators will plan for 54 patients (approximately 27 per study arm). The investigators performed similar calculations for the consent rate outcome using a feasibility threshold of 75% and an expected consent rate of 90% leading to an identical sample size number.

KANINE Pilot Study Analysis Calculation of the 3 feasibility outcomes for the KANINE trial are noted in the outcomes section above. The analysis and reporting of results will follow the CONSORT guidelines for reporting of randomized pilot and feasibility trials25. The process of participant enrolment and flow throughout the study will be summarized using a flow-diagram. Participant demographics, medical history, and secondary outcomes will be summarized by treatment group using descriptive summary measures: expressed as mean and standard deviation or median and interquartile range for continuous variables, depending on the distribution, and number and percent for binary/categorical variables.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years) admitted to the ICU
* Receiving invasive mechanical ventilation and expected to remain mechanically ventilated beyond the calendar day after randomization
* Mechanically ventilated for fewer than 3 days
* Receiving any non-ketamine continuous sedative infusion

Exclusion Criteria:

* Admitted with a primary diagnosis of intracranial hemorrhage, traumatic brain injury, or stroke
* Admitted with uncontrolled hypertension (SBP/DBP > 180/100mmHg)
* Status asthmaticus
* Admitted to the ICU with partial thickness burns > 10% total body surface area or any full thickness burns
* Schizophrenia
* End-stage Liver Failure (Child-Pugh C)
* Requiring an equivalent of norepinephrine at a dose ≥1mcg/kg/min
* Undergoing palliation or comfort care
* On neuromuscular blocking agent
* Pre-existing tracheostomy
* Hypersensitivity to Ketamine
* Liver transplantation in the last month
* Pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Recruitment Rate | 3 months
  Feasibility will be judged by the 3 outcomes of recruitment rate, consent rate, and protocol adherence. We define a successful recruitment rate of 0.5 patients per centre per month over the duration of the trial.
Feasibility: Consent Rate | 3 months
  This will be judged by the 3 outcomes of recruitment rate, consent rate, and protocol adherence. We will define >75% consent rate as successful.
Feasibility: Protocol Adherence | 3 months
  This will be judged by the 3 outcomes of recruitment rate, consent rate, and protocol adherence. We will define ≥75% protocol adherence as successful.

SECONDARY OUTCOMES:
Ventilator-free Days at 28 days | 28 Days
28-day mortality | 28 Days
ICU Mortality | 3 months
ICU Length of Stay | 3 months
Number of Participants receiving a Tracheostomy | 3 months
Hospital Mortality | 3 months
Hospital Length of Stay | 3 months
Delirium | 28 Days
  Delirium will be reported using the validated Confusion Assessment Method for the ICU (CAM-ICU) score (dichotomous score) or the Intensive Care Delirium Screening Checlist (ICDSC).
  Minimum Value: No Delirium Maximum Value: Delirium
Delirium-Free/Coma-Free Days at 14 days | 14 days
Use of anti-psychotics (total dosage) | 28 Days
Use of benzodiazepines (total dosage) | 28 Days
Post-traumatic stress disorder symptoms at 3 months post ICU discharge | 3 months
  This outcome will use the validated Impact of Event Scale - Revised
  Minimum Value: 0 Maximum Value: 88
  Value ≥ 33 consistent with PTSD
Total dosage of continuous sedative requirements over ICU stay | 28 Days
  This outcome will report the total dosage and weight-based mean dosage of continuous sedatives used in the ICU
Total dosage of analgesic requirements over ICU stay | 28 Days
  This outcome will report the total dosage and weight-based mean dosage of analgesics used in the ICU
Number of participants with arrhythmias | 28 Days
  Inclusive of atrial flutter/fibrillation, ventricular fibrillation, ventricular tachycardia
Number of times participants have emesis/vomiting | 28 Days
  Reported incidents of vomiting.

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Hamilton Health Sciences, Hamilton, Ontario
  - Mount Sinai Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
The results of this study will be submitted for publication in a medical journal. In the future, we may use our individual patient data ourselves to conduct a meta-analysis with our own team.